CLINICAL TRIAL: NCT03299725
Title: A Prospective Open-label Study on Efficacy and Tolerability of Colloidal Bismuth Sub-citrate as Adjunctive Therapy to a Combination of Esomeprazole, Amoxicillin and Metronidazole for 10 Days for Helicobacter Pylori Elimination in Children
Brief Title: Bismuth Based Quadruple Therapy 10 Days in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBS-EAM 10d
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: colloidal bismuth sub-citrate

INTERVENTIONS:
Drug: colloidal bismuth sub-citrate — colloidal bismuth sub-citrate administered as an adjunctive therapy in combination with esomeprazole, amoxicillin and metronidazole

SUMMARY:
Helicobacter pylori infection causes chronic gastritis, peptic ulcer disease and is involved in the development of gastric cancer.

Current accepted strategies to eliminate the infection in children are a 10 days sequential treatment (proton pump inhibitor + amoxicillin 5 days followed by proton pump inhibitor + metronidazole + clarithromycin 5 days) or a triple therapy 14 days (proton pump inhibitor + amoxicillin + clarithromycin or metronidazole).

However, there is a concern due to the growing resistance of Helicobacter pylori strains to antibiotics, especially clarithromycin, and the decreased efficacy of first line treatment regimens to satisfactorily eliminate the infection in children.

Recent data show that combinations using bismuth salts must be considered in adults. Indeed, the efficacy of a 10 days of quadruple therapy with omeprazole plus a single three-in-one capsule containing bismuth subcitrate, metronidazole and tetracycline was shown to be highly superior to the standard triple therapy combining omeprazole, amoxicillin, and clarithromycin without related severe adverse events.

The possibility of re-using bismuth salts on a more regular basis in pediatrics is being restudied through a monocentric, prospective, open label, single arm clinical trial to assess the safety and efficacy of a 10 days colloidal bismuth sub-citrate as an adjunctive therapy in combination with esomeprazole, amoxicillin and metronidazole in children aged 6-17 years, infected by Helicobacter pylori.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric subjects aged 6 to 17 years of either gender
* Body weight ≥ 20kg.
* Helicobacter pylori gastritis confirmed by positive histology and culture with antimicrobial susceptibility testing.
* Antral and corpus biopsies must have been taken for histology and culture during an upper GI endoscopy performed for chronic or recurrent pain in the epigastric region with epigastric tenderness at physical examination.
* Subject able to swallow tablets.
* All girls of child-bearing potential must have a negative urine pregnancy test at Visit 1. If sexually active, girls of child-bearing potential and boys whose partner is of child-bearing potential agree to use highly effective method of birth control during the trial.
* In the Investigator's opinion, patient is willing and able to comply with all trial requirements specified in this protocol.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.
* Subjects (or their legally-acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study. Assent is also required of children capable of understanding the nature of the study (typically older than 11 years of age).

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Have a history of significant renal or hepatic impairment.
* Have an erosive esophagitis or peptic ulcer disease in the gastric or the duodenal mucosa showed during the upper GI endoscopy.
* Have received proton pump inhibitors within 2 weeks prior to first administration of study agent.
* Have received any antimicrobial agent within 4 weeks prior to first administration of study agent.
* Require routine use (≥ 2 times per week) of non-steroidal anti-inflammatory drug (NSAID).
* Are under any immunosuppressive agent.
* Are under oral or IV steroids
* Have a scheduled elective surgery or any procedures requiring general anaesthesia during the trial.
* Have known allergies or a known hypersensitivity to any Study Drugs or their excipients (refer to Study Drugs SmPCs).
* Contraindication for any of the Study Drugs (refer to Study Drugs SmPCs).
* Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.
* Subjects who are participating or have participated in another study with an IMP in the past 12 weeks.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-11-24 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
13C-urea breath test | Week 10
  Ratio of 13C/12C, expressed as delta 13C in pro mil, and compared with PeeDee Belemnite calcium carbonate standard

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse event | Up to 10 weeks after start of study treatment
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Adherence to the study treatment | week 2
  Adherence reported by patient on a diary card and study drug accountability
Intestinal microbiome analysis | Week 0
  Qualitative description
Intestinal microbiome analysis | Week 10
  Changes in the relative phylum-level abundance in the stools, based on 16S rRNA classification, between week 0 and week 10
Effect of antimicrobial resistance on the success rate | Week 10
  Qualitative description

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Kanfaoui, MD, Study Director — Queen Fabiola Children's University Hospital
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No